CLINICAL TRIAL: NCT03413566
Title: Trends in Prevalence and Comorbidities of Children With Cerebral Palsy in Norway Born 1996 to 2010
Brief Title: Trends in Prevalence and Comorbidities of Children With Cerebral Palsy in Norway
Status: Enrolling by invitation | Type: Observational
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Norwegian University of Science and Technology (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Guro L. Andersen, Senior Consultant, Leader of the Cerebral Palsy Registry of Norway, Sykehuset i Vestfold HF
Other Study IDs: 197590
Record Dates: First submitted 2018-01-04; First posted 2018-01-29 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Cerebral Palsy
Keywords: Trends; Prevalence; Registries/statistics & numerical data; Epidemiology
MeSH Terms: conditions — Cerebral Palsy | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with clinical diagnosis of CP: All children residing in Norway with a validated diagnosis of cerebral palsy.
  Interventions: Other: Clinical diagnosis
- Children without CP: All children residing in Norway without a diagnosis of cerebral palsy.

INTERVENTIONS:
Other: Clinical diagnosis — A clinical diagnosis of cerebral palsy given by a pediatrician at a habilitation center in Norway.
  Groups: Children with clinical diagnosis of CP

SUMMARY:
Many studies have reported that the prevalence of cerebral palsy (CP) has been relatively stable and is mainly due to events before birth and therefore cannot be prevented. However, these studies were undertaken in populations born towards the end of the last century. There has since been significant improvement in both obstetrical and neonatal intensive care.

The main aim is to investigate trends in the prevalence and clinical characteristics of children with CP in Norway born from 1996 to 2010 in order to gain a modern understanding of the panorama of CP in Norway. The investigators suspect that improved methods of obstetrical and neonatal care introduced in Norway during the last 20 years has resulted in a decrease in the prevalence of CP as well as in the proportion of children with severe CP subtypes and comorbidities. The long term aim is to improve the quality of pregnancy care and newborn medicine for children at risk of CP, and to ensure equal diagnostics and treatment of patients with CP, regardless of place of residence in Norway.

For this project, the investigators will use data from three national health registers: The Cerebral Palsy Registry of Norway (CPRN), The Medical Birth Registry of Norway and The Norwegian Patient Registry (NPR). The use of data from these high quality health registries provides us with a unique opportunity to study our aims on a population level, as well as per health region/health trust.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of permanent motor disabilities in children, and one of the patient groups that receive the largest proportion of health care resources in high-income countries. CP is the result of a non-progressive injury in the immature brain that occurs before, during or after birth (neonatal period). The injury may be caused by a congenital brain abnormality, infection, trauma or other complications. Known risk factors include premature birth, restricted fetal growth and lack of oxygen during birth (birth asphyxia). Research shows that the panorama of causes has changed over time.

The clinical characteristics of CP vary considerably, something one would expect from the variation in potential causes. CP is categorized into subtypes based on the dominating symptoms and which part of the body is affected. Further classification is often based on the severity of the child's motor impairment. Also, children with CP often have additional comorbidities such as epilepsy, impaired vision and/or hearing, impaired ability to speak/communicate, cognitive disorders, and nutritional problems. Nor in these areas has the situation remained static over time.

During the last 20 years, both obstetric and neonatal care has undergone significant changes in Norway as well as in other countries. In the 1990s surfactant treatment of premature children was established, and in the early 2000s, therapeutic hypothermia was introduced as a new treatment for term born children with hypoxic ischemic encephalopathy (HIE). There have also been improvements in fetal monitoring during labor from around 2004 with an increase in the use of continuous electronic monitoring of the fetal heart using either the cardiotocography (CTG) or ST analysis (STAN) method to assess the baby's well-being, as well as Fetal scalp pH testing to determine if the baby is getting adequate oxygen supply. In this project, the investigators intend to study if the introduction of these new treatments has been associated with a decrease in the prevalence of CP and in changes in the clinical picture (e.g. less serious motor disabilities and comorbidities) for children born 1996 to 2010.

To study these questions, the investigators will take advantage of data from three national health registers: The Medical Birth Registry of Norway (MBRN), The Norwegian Patient Registry (NPR) and The Cerebral Palsy Registry of Norway (CPRN). While the MBRN has recorded all births since 1967, the NPR has recorded all patients treated in special health care service since 1997 and with their national identification numbers since 2008. All children with CP are diagnosed and their treatment assessed at pediatric habilitation centers, reporting to the NPR. The CPRN is a national medical quality register, owned by the South-Eastern Norway Regional Health Authority, and is located at the Vestfold Hospital Trust. Participation in the CPRN is based-on parental informed consent. This register has systematically recorded children with CP born since 1996, and has received high scores by The Norwegian Advisory Unit for Medical Quality Registries (SKDE). Moreover, the investigators have recently documented completeness and correctness of CP diagnoses in the CPRN as well as in the NPR. Thus, the use of data from these three high quality health registries provides a unique opportunity to study on a population level if the new obstetric and neonatal treatment options have been followed by measurable reductions in the prevalence of CP.

The purpose of the Cerebral Palsy Registry of Norway is to increase knowledge of the causes and treatment of children and youths with CP through surveillance and systematic analyses, including to:

* Describe the prevalence of CP in Norway, including subtypes, severity and comorbidities
* Improve the quality of pregnancy care and newborn medicine
* Ensure equal treatment and follow-up of children/youths with CP in Norway, regardless of place of residence.
* Increase knowledge of CP

This study fulfills all of these aims, and also has the potential to go one step further and impact children at risk for CP. By gaining better knowledge of children with CP in Norway during this study period, the investigators can explore variations in the causes and treatments for newborns at increased risk of CP and children with CP, per health region and/or per health trust.

The overall design of this project is a register-based population study, comprising of three sub-studies.

Study 1: Completeness and correctness of the CPRN and NPR There was a variation in the reported prevalence of CP in Norway from different data sources used to identify children with CP. The aim of this study was thus to combine data sources and to validate the CP population in Norway for children born 1996-2007, and thereby gain an accurate estimate of the prevalence rate of CP in Norway. This study was published in March 2017. A second validation study of CP diagnoses for children born 2007-2010 and registered in the CPRN and/or NPR was completed in January 2017.

Study 2: Trends in prevalence, causes, diagnostics and clinical characteristics of children with cerebral palsy born in Norway 1999 to 2010.

The aim of this study will be to examine whether there has been a decrease in the prevalence of CP and changes in the clinical picture (e.g. less serious motor disabilities and comorbidities) following new standardized methods of obstetrical care, such as fetal monitoring during labor, as well as of intensive care of sick newborns introduced in Norway during the last 20 years.

Data for 707 916 children born in Norway between 1999 and 2010 have been registered in the MBRN. Of these, 1664 children have been confirmed to have CP and are registered in the CPRN. A data linkage of the MBRN and CPRN was performed in February 2017. The MBRN includes data on a number of well-known and unknown risk factors for CP (e.g. length of pregnancy, Apgar scores, congenital malformations, intrauterine growth retardation, etc.). The CPRN contains information on the clinical picture of CP at five years of age (gross, fine and oral motor function, cognition, epilepsy, eating abilities, and magnetic resonance imaging findings).

Logistic regression using fractional polynomials will be used to estimate time trends in prevalence rates with 95% confidence intervals (CI), according to Altman et al. Differences in proportions of clinical characteristics will be analyzed by χ2 linear-by-linear association or Cochran-Armitage test for trends. A p-value below 0.05 is considered statistically significant.

Data analysis began in early 2017, and an article is currently being finalized.

Study 3: CP and comorbidities Data from the NPR will be used, including administrative (treating institution, consultation and/or hospitalization, patient place of residence) and medical (diagnosis and treatments codes) and social (housing situation and care situation) data on all children born 1996-2010 that have received treatment in specialist health services since 2008. Children with CP will be compared to children without a CP diagnosis. The main aim of this study will be to describe frequencies of comorbidities that occurred before and after children are diagnosed with CP. Logistic regression analyses will be used to compare children with CP to the general population. This study is a follow-up study in collaboration with the Norwegian National Institute of Public Health, which recently published a study on Comorbidity and Childhood Epilepsy: A Nationwide Registry Study.

ELIGIBILITY:
Inclusion Criteria:

* Validated diagnosis of cerebral palsy

Exclusion Criteria:

* No diagnosis of cerebral palsy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children residing in Norway born from 1996 to 2010 with a diagnosis of cerebral palsy, confirmed by a pediatrician at one of the habilitation centers in the country.
Sampling Method: Non-Probability Sample
Enrollment: 707916 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cerebral palsy | Registration at 5 years of age
  Assessment of number of children with cerebral palsy per 1000 live births
Prevalence of cerebral palsy subtypes | Registration at 5 years of age
  Assessment of cerebral palsy severity according to Surveillance of Cerebral Palsy in Europe classification tree of CP subtypes: spastic unilateral, spastic bilateral, dyskinetic, ataxic and mixed/unspecified, per 1000 live births

SECONDARY OUTCOMES:
Gross Motor Function Classification System (GMFCS) | Registration at 5 years of age
  Assessment of motor function severity on five levels. I: Walks without limitations. II: Walks with limitations. III: Walks using a hand-held mobility device. IV: Self-mobility with limitations; may use powered mobility. V: Transported in a manual wheelchair.
Epilepsy | Registration at 5 years of age
  Assessment of epilepsy according to Surveillance of Cerebral Palsy in Europe guidelines on two levels. I: present. II: not present.
Cognition | Registration at 5 years of age
  Assessment of cognitive abilities according to Surveillance of Cerebral Palsy in Europe on two levels. I: normal (IQ test score above 70 or clinically assessed). II: intellectual disability (IQ test score below 70 or clinically assessed).
Viking Speech Scale | Registration at 5 years of age
  Assessment of speech production on four levels. I: Speech is not affected by motor disorder. II: Speech is imprecise but usually understandable to unfamiliar listeners. III: Speech is unclear and not usually understandable to unfamiliar listeners out of context. IV: No understandable speech.
Eating and Drinking Ability Classification System (EDACS) | Registration at 5 years of age
  Assessment of eating ability on five levels. I: Eats and drinks safely and efficiently. II: Eats and drinks safely but with some limitations to efficiency. III: Eats and drinks with some limitations to safety; maybe limitations to efficiency. IV: Eats and drinks with significant limitations to safety. Level V: Unable to eat or drink safely - tube feeding may be considered to provide nutrition.
Visual impairment | Registration at 5 years of age
  Assessment of visual function according to Surveillance of Cerebral Palsy in Europe guidelines on three levels. I: normal. II: impaired. III: severely impaired (blind i.e. <6/60 (<0·1) before correction on the best eye)
Hearing impairment | Registration at 5 years of age
  Assessment of hearing ability according to Surveillance of Cerebral Palsy in Europe guidelines on three levels. I: normal. II: impaired. III: severely impaired (loss > 70 dB before correction on the best ear).
Other medical and psychiatric conditions - International Statistical Classification of Diseases and Related Health Problems 10th revision codes (ICD-10) | Registration at 5 years of age
  Assessment of frequencies of other medical and psychiatric conditions according to ICD-10 diagnosis codes.

CONTACTS AND LOCATIONS:
Overall Officials: Guro L Andersen, MD, PhD, Principal Investigator — Vestfold Hospital Trust/The Cerebral Palsy Registry of Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available due to national medical quality registry status and Norwegian data protection laws.

REFERENCES:
- [Result] Hollung SJ, Vik T, Wiik R, Bakken IJ, Andersen GL. Completeness and correctness of cerebral palsy diagnoses in two health registers: implications for estimating prevalence. Dev Med Child Neurol. 2017 Apr;59(4):402-406. doi: 10.1111/dmcn.13341. Epub 2016 Nov 29. PMID 27896812
- [Result] Hollung SJ, Vik T, Lydersen S, Bakken IJ, Andersen GL. Decreasing prevalence and severity of cerebral palsy in Norway among children born 1999 to 2010 concomitant with improvements in perinatal health. Eur J Paediatr Neurol. 2018 Sep;22(5):814-821. doi: 10.1016/j.ejpn.2018.05.001. Epub 2018 May 8. PMID 29779984